CLINICAL TRIAL: NCT04839692
Title: Assessment and Augmentation of Lip Appearance in Specific Study Populations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dieter Manstein, MD (Other)
Responsible Party: Sponsor-Investigator, Dieter Manstein, MD, Principal Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021P000010
Record Dates: First submitted 2021-02-25; First posted 2021-04-09 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Lip Aging; Lip Augmentation; Lip
MeSH Terms: conditions — Lymphoid Interstitial Pneumonia

STUDY DESIGN:
Intervention Model Description: Investigators will enroll 40 subjects; 20 subjects who are 21-30 years old and 20 subjects who are post-menopausal women. Both groups will receive identical treatments.
Who Masked: Investigator
Masking Description: Standard photographs will be blindly reviewed by a physician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Young females (21-30 years old) (Other): young healthy females (21-30 years old) from all phototypes who have thin or moderately thick lips
  Interventions: Drug: Hyaluronic acid filler
- post menopausal females (Other): post menopausal females from all phototypes who have thin or moderately thick lips
  Interventions: Drug: Hyaluronic acid filler

INTERVENTIONS:
Drug: Hyaluronic acid filler — Hyaluronic acid filler treatment of the lips with Restylane Kysse, which is a FDA approved treatment for lip augmentation.

SUMMARY:
This study aims to learn more about the effects of aging and lip filler treatment on lips and the surrounding skin by comparing, among two different age groups of people, changes in the blood vessels and nerves, volume, color and texture change before and after lip filler treatment and pain tolerance from lip filler treatment.

DETAILED DESCRIPTION:
This study will investigate aging of the cutaneous changes of human skin anatomy in the lips and perioral area to better understand and quantify the aging process in this, including the effect of age on lip redness. Additionally, the investigators aim to test the effects of a common lip augmentation procedure, hyaluronic-acid based fillers, on the appearance (volume, texture and color) of aging lips, in addition to the tolerability of this procedure. It is hypothesized that dermal lip fillers may decrease the redness of the lips.

Besides, the investigators want to evaluate oxytocin level changes and relate it to subjects' satisfaction after the lip filler procedure.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be able and willing to provide written informed consent and comply with the requirements of the study protocol;
* In good general health, based on answers provided during the screening visit;
* Subjects must be able to read and understand English;
* Caucasian female;
* Aged 21-30 years and post-menopausal;
* Skin Types (all Fitzpatrick Skin Phototypes );

  * Smoking history is self-report.
* Have very thin to moderately thick lips (Lip Fullness Grading Scale [LFGS] scores 0-2).

Exclusion Criteria:

* Participation in another investigational drug or device clinical trial in the past 30 days;
* Are pregnant or lactating;
* Intake of hormone replacement therapy (HRT) in the past 6 months;
* Have a history of drug or alcohol abuse or have reported habitual alcohol intake greater than 2 standard drinks per day [e.g., 2 beers, 2 glasses of wine, or 2 mixed drinks];
* Presence of eczema, psoriasis, or any other skin disease on the lips or perioral skin;
* Have birth marks, tattoos, scars, or any other disfiguration of the skin in the skin area of interest;
* Use of any anti-aging skin care products containing retinoic acid, retinol, or other retinoids (e.g. tazarotene, adapalene) or estrogen on the skin area of interest in the past 6 months;
* Use of any prescription topical medication, such as corticosteroids or hydroquinone on the skin area of interest in the past 6 months;
* Have a history of photodynamic therapy treatment or any skin rejuvenation procedure on the skin area of interest;
* History of blood-clotting abnormality;
* History of keloid formation or hypertrophic scarring;
* Clinically significant abnormal findings or conditions which might, in the opinion of the Investigator, interfere with study evaluations or pose a risk to subject safety during the study;
* Exhibits any clinical conditions or takes any medication which in the opinion of the investigator may interfere with the study or pose a risk to subject safety during the study;
* Is not able to follow study protocol;
* Have permanent lip implant, and lip enhancement or laser therapy performed within the preceding 12 months;
* Known history of allergy or sensitivity to glycerol, Tegaderm, lidocaine, hyaluronic acid dermal fillers or materials with gram-positive bacterial proteins.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-05-07 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Manstein, MD, PhD, Principal Investigator — Massachusetts General Hospital; Neera Nathan, MD, MSHS, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH Clinical Unit for Research Trials & Outcomes Research, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers.

REFERENCES:
- [Background] Uitto J. Understanding premature skin aging. N Engl J Med. 1997 Nov 13;337(20):1463-5. doi: 10.1056/NEJM199711133372011. No abstract available. PMID 9358147
- [Background] Zouboulis ChC. [Intrinsic skin aging. A critical appraisal of the role of hormones]. Hautarzt. 2003 Sep;54(9):825-32. doi: 10.1007/s00105-003-0581-7. German. PMID 12955259
- [Background] Leung WC, Harvey I. Is skin ageing in the elderly caused by sun exposure or smoking? Br J Dermatol. 2002 Dec;147(6):1187-91. doi: 10.1046/j.1365-2133.2002.04991.x. PMID 12452869
- [Background] Argyropoulos AJ, Robichaud P, Balimunkwe RM, Fisher GJ, Hammerberg C, Yan Y, Quan T. Alterations of Dermal Connective Tissue Collagen in Diabetes: Molecular Basis of Aged-Appearing Skin. PLoS One. 2016 Apr 22;11(4):e0153806. doi: 10.1371/journal.pone.0153806. eCollection 2016. PMID 27104752
- [Background] van Waateringe RP, Mook-Kanamori MJ, Slagter SN, van der Klauw MM, van Vliet-Ostaptchouk JV, Graaff R, Lutgers HL, Suhre K, El-Din Selim MM, Mook-Kanamori DO, Wolffenbuttel BHR. The association between various smoking behaviors, cotinine biomarkers and skin autofluorescence, a marker for advanced glycation end product accumulation. PLoS One. 2017 Jun 20;12(6):e0179330. doi: 10.1371/journal.pone.0179330. eCollection 2017. PMID 28632785
- [Background] Gilchrest BA, Soter NA, Hawk JL, Barr RM, Black AK, Hensby CN, Mallet AI, Greaves MW, Parrish JA. Histologic changes associated with ultraviolet A--induced erythema in normal human skin. J Am Acad Dermatol. 1983 Aug;9(2):213-9. doi: 10.1016/s0190-9622(83)70131-3. PMID 6886112
- [Background] Rogers GS, Gilchrest BA. The senile epidermis: environmental influences on skin ageing and cutaneous carcinogenesis. Br J Dermatol. 1990 Apr;122 Suppl 35:55-60. doi: 10.1111/j.1365-2133.1990.tb16126.x. PMID 2186787
- [Background] Bentov I, Reed MJ. The effect of aging on the cutaneous microvasculature. Microvasc Res. 2015 Jul;100:25-31. doi: 10.1016/j.mvr.2015.04.004. Epub 2015 Apr 24. PMID 25917013
- [Background] Tamura E, Ishikawa J, Sugata K, Tsukahara K, Yasumori H, Yamamoto T. Age-related differences in the functional properties of lips compared with skin. Skin Res Technol. 2018 Aug;24(3):472-478. doi: 10.1111/srt.12456. Epub 2018 Feb 6. PMID 29405429
- [Background] Hilton S, Sattler G, Berg AK, Samuelson U, Wong C. Randomized, Evaluator-Blinded Study Comparing Safety and Effect of Two Hyaluronic Acid Gels for Lips Enhancement. Dermatol Surg. 2018 Feb;44(2):261-269. doi: 10.1097/DSS.0000000000001282. PMID 29059146
- [Background] Stojanovic L, Majdic N. Effectiveness and safety of hyaluronic acid fillers used to enhance overall lip fullness: A systematic review of clinical studies. J Cosmet Dermatol. 2019 Apr;18(2):436-443. doi: 10.1111/jocd.12861. Epub 2019 Jan 12. PMID 30636365
- [Background] Savoia A, Accardo C, Vannini F, Di Pasquale B, Baldi A. Outcomes in thread lift for facial rejuvenation: a study performed with happy lift revitalizing. Dermatol Ther (Heidelb). 2014 Jun;4(1):103-14. doi: 10.1007/s13555-014-0041-6. Epub 2014 Jan 17. PMID 24436079
- [Background] Carruthers A, Carruthers J, Hardas B, Kaur M, Goertelmeyer R, Jones D, Rzany B, Cohen J, Kerscher M, Flynn TC, Maas C, Sattler G, Gebauer A, Pooth R, McClure K, Simone-Korbel U, Buchner L. A validated lip fullness grading scale. Dermatol Surg. 2008 Nov;34 Suppl 2:S161-6. doi: 10.1111/j.1524-4725.2008.34365.x. PMID 19021674
- See also: Restylane Kysse Patient Brochure — https://www.galderma.com/us/sites/g/files/jcdfhc341/files/2020-04/Restylane_Kysse-Patient_Brochure.pdf?_ga=2.59052845.1698235642.1604334264-853585669.1604334264&_gac=1.157524424.1604378565.CjwKCAiA-f78BRBbEiwATKRRBPyH8_64L0BLjGEHNISljih9I6tz-fSQohCtDMdwKAe7hz57dYQAihoCieQQAvD_BwE

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Young Females (21-30 Years Old) | Post Menopausal Females
Started | 23 | 14
Completed | 22 | 11
Not Completed | 1 | 3
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Young Females (21-30 Years Old) | Post Menopausal Females | Total
Number analyzed (Participants) | 22 | 11 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 5 | 27
  >=65 years | 0 | 6 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.72 (2.64) | 69.91 (10.97) | 39.79 (22.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 11 | 33
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 21 | 9 | 30
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 11 | 33

OUTCOME MEASURES:

1. Primary Outcome: Change in Lip Vessel's Thickness
Description: Pre and post-treatment lip vessel thickness was measured in µm using Optical Coherence Tomography-Angiography imaging. For each age group, pre and post-treatment means were calculated.
  The difference between the post and the pre-treatment means is shown below (post-treatment mean - pre-treatment mean).
Time Frame: Day 1 and Day 14
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Young Females (21-30 Years Old) | Post Menopausal Females
Number analyzed (Participants) | 22 | 11
µm | 0.833 (1.334) | 0.360 (1.543)

2. Secondary Outcome: Wong-Baker FACES Pain Rating Scale
Description: This scale will be used to record the subject's overall pain from the procedure. There are 6 faces ranging from 0=no pain to 10=the worst pain.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Young Females (21-30 Years Old) | Post Menopausal Females
Number analyzed (Participants) | 22 | 11
score on a scale | 2.9 (.5) | 3.5 (0.14)

3. Secondary Outcome: Lip Fullness Measurement (Measures the Increase of Lip's Size After the Procedure)
Description: The Lip Fullness Grading Scale was used to measure the size of the lips before and after the procedure in both groups. The result presented below is the difference between the means after and before the procedures for each group.
  min value: 0 - very thin lips - worse outcome Max value: 4 - full lips- a better outcome
Time Frame: D1 and D14
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Young Females (21-30 Years Old) | Post Menopausal Females
Number analyzed (Participants) | 22 | 11
units on a scale | 1.14 (0.52) | 0.78 (0.34)

ADVERSE EVENTS:
Time Frame: 21 days
Description: Minimal-risk study with healthy participants. Two subjects from the young arm presented lip asymmetry as an adverse event.
Arm/Group | Young Females (21-30 Years Old) | Post Menopausal Females
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/11
Other Adverse Events (participants affected / at risk) | 2/22 | 0/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Young Females (21-30 Years Old) (N=22) | Post Menopausal Females (N=11)
Asymmetry (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) — Asymmetry of lips

LIMITATIONS AND CAVEATS:
Smaller number of subjects in postmenopausal group due to the difficulties in recruitment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-29): https://cdn.clinicaltrials.gov/large-docs/92/NCT04839692/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT04839692/ICF_001.pdf